CLINICAL TRIAL: NCT05170503
Title: Neoadjuvant Sintilimab Plus SOX in the Locally Advanced Esophagogastric Junction Adenocarcinoma: a Prospective, Single Arm Phase II Trial
Brief Title: Neoadjuvant Immunochemotherapy in Locally Advanced Esophagogastric Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yang Hong, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC B2021-356-01
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Esophagogastric Junction Adenocarcinoma
Keywords: Esophagogastric Junction Adenocarcinoma; neoadjuvant; chemo-immunotherapy; Sintilimab
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant chemo-immunotherapy (Experimental): Neoadjuvant Immunotherapy (Sintilimab, PD-1 inhibitor) Combined With Chemotherapy (Tegafur+Oxaliplatin) Each patient will complete 3 cycles of neoadjuvant therapy. After evaluating the radiographical response, operation with curative extent (Ivor-lewis or Mckeown procedure with two-field lymph node dissection) will be performed after 6 to 8 weeks from the last cycle of neoadjuvant treatment. Patients with and without surgery enter the survival follow-up period.
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg iv drip. Qd D1 + Oxaliplatin 130/m2 iv drip. Qd D1 + Tegafur (Gimeracil and Oteracil Potassium Capsules) [40mg/m2 if BSA <1.25m2, 50mg/m2 if BSA ≥1.25m2 & <1.5m2, 60mg/m2 if BSA ≥1.5m2] po. Bid D1-14 for three cycles

SUMMARY:
The purpose of this study is to access the safety and efficacy of neoadjuvant Immunotherapy (Sintilimab, PD-1 inhibitor) combined with chemotherapy (Tegafur+Oxaliplatin) for locally advanced esophagogastric junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced esophagogastric junction Adenocarcinoma cT3-4aN0 or T1-4aN1-3M0
* No previous anti-tumor treatment
* ECOG PS: 0-1
* The functions of important organs meet the following requirements (excluding the use of any blood components and cell growth factors during the screening period)：Absolute neutrophil count ≥ 1.5 × 109/L； Platelet ≥ 90 × 109/L； Hemoglobin ≥ 9g / dl; Serum albumin ≥ 3G / dl; Thyroid stimulating hormone (TSH) ≤ ULN (if abnormal, the levels of T3 and T4 should be investigated at the same time. If the levels of T3 and T4 are normal, they can be included in the group); Bilirubin ≤ ULN; ALT and AST ≤ 1.5 times ULN; AKP ≤ 2.5 times ULN; Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60ml / min.
* Women of childbearing age must have taken reliable contraceptive measures or conducted pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and are willing to use appropriate contraceptive methods during the test and 8 weeks after the last administration of test drugs. For men, they must agree to use appropriate methods of contraception or surgical sterilization during the trial and 8 weeks after the last administration of the trial drug.
* The patients voluntarily joined the study and signed the informed consent form. They had good compliance and cooperated with the follow-up.

Exclusion Criteria:

* Known Her-2 positive
* Any active autoimmune disease or history of autoimmunity (as follows, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism and hypothyroidism; Subjects with vitiligo or asthma in childhood have been completely relieved and do not need any intervention after adulthood can be included; Asthma in which subjects need bronchodilators for medical intervention cannot be included).
* Severe allergic reaction to monoclonal antibody.
* The number of neutrophils in peripheral blood was less than 1500 / mm3.
* There are cardiac clinical symptoms or diseases that are not well controlled.
* Previously received radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeted therapy.
* The subjects were innate or acquired immunodeficiency (such as HIV), or active hepatitis (hepatitis B reference: HBsAg) positive, HBVDNA > 2000IU/ml or copy number > 104/ml; Hepatitis C reference: HCV antibody positive.
* According to the judgment of the researcher, the subject has other factors that may lead to the forced midway termination of this study, such as other serious diseases (including mental diseases) requiring combined treatment, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subject, or the collection of data and samples.
* The researchers judged the patients with high risk of esophageal perforation or no potential possibility of surgery through endoscopic ultrasonography or imaging.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | From date of enrollment until one month after resection
  No malignant tumor cells were detected in the removed specimens including primary tumor and lymph nodes

SECONDARY OUTCOMES:
Overall survival | 2-5 years
  The time from randomization to death from any cause.
Disease-Free-Survival | 2-5 years
  The time between the beginning of treatment and the observation of disease progression or death from any cause.
R0 resection rate | From date of enrollment until one month after resection
  The percentage of patients who undergo complete resection

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
upon reaseonable request with a plan